CLINICAL TRIAL: NCT05499559
Title: Digitally Delivered Education and Exercises for Patients With Hand Osteoarthritis-An Observational Study
Brief Title: Effects of 12-week Digital Treatment in Patients With Hand OA on Pain and Function
Status: Completed | Type: Observational
Sponsor: Joint Academy (Industry)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: HandOA2022
Record Dates: First submitted 2022-08-02; First posted 2022-08-12 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Hand Osteoarthritis; Wrist Osteoarthritis; Thumb Osteoarthritis; Finger Osteoarthritis
Keywords: Telemedicine; Telehealth; Mobile Health; eHealth; mHealth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Joint Academy: The participants receive the digital treatment of Joint Academy.
  Interventions: Behavioral: Joint Academy digital treatment

INTERVENTIONS:
Behavioral: Joint Academy digital treatment — The Joint Academy® (www.jointacademy.com) program for people with hand OA consists of video instructed and progressively adaptable daily exercises, patient education through text lessons, possibility for a social chat group with other patients and a continuous asynchronous chat function with a personal reg. physiotherapist who supervises the patient during the full participation period. The program also contains three telephone consultations with a physiotherapist that were compulsory, one at the start, one after six weeks and one after three months.

SUMMARY:
The purpose of this study is to evaluate the effect of a 12 week digital treatment program for patients with hand osteoarthritis. The treatment consisted of exercises and educational sessions with respect to the disease, its natural course and recommended treatment strategies.

Design: An observational longitudinal cohort study.

The investigators will include participants who participated in the digital treatment of Joint Academy® for 3 months.

Outcomes: Investigators will analyze pain with Numeric Rating Scale (NRS) 0-10 (best to worst), function with the Functional Index for Hand OsteoArthritis (FIHOA) and health related quality of life with EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) at baseline and at 3 months. Main outcome will be change in pain. The investigators will also analyze minimally clinical important changes (improved or not) and mean changes in EQ-5D-5L index score, pain and function.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of the leading causes of disability worldwide and due to its rising prevalence, the identification of appropriate care and care delivery modalities is a priority for the health care systems. Exercise and education constitute the first-line intervention for people with knee, hip and hand OA and have been shown to be effective regardless of symptoms and disease severity. International guidelines recommend that first-line interventions for the majority of musculoskeletal conditions should involve nonsurgical management with exercise and education guided by a physiotherapist (PT) and based on a personalised care approach.

OA of the hand is probably the most common form of OA and almost 50% of women and 25% of men will be affected during the life course. Self-management strategies includes a wide range of strategies such as education for strengthening or stretching exercises, joint protection education for activity and pacing, use of proper body mechanics, and assistive devices to improve pain, reduce inflammation, lower additional risk of deformities, and enhance performance. Systematic reviews that compared joint protection strategies to usual care have shown similar effects at short-term and superior effects at mid- and long-term compared to usual care.

To implement the guidelines, the Better Management of Patients with OsteoArthritis (BOA), a face-to-face concept including education and an option to exercise, has been developed and is offered at primary care clinics in Sweden since 2008 for patients with hip- knee- and hand OA. BOA has previously been found to reduce pain and improve function and quality of life in patients with hip and knee OA. Unfortunately, there is a discrepancy between recommended treatment and what patients receive and around 30% of people with OA seeking care go through first line management.

Traditional face-to-face interventions present barriers, such as limited access and lack of flexibility, which may limit the patients' adherence with the interventions. Digital delivery of the management program may be one way of overcoming such barriers. Telehealth, defined as the 'delivery of healthcare at a distance using information and communication technology' could be a solution to many access barriers and has been rapidly adopted by many healthcare professions and accelerating even more throughout the COVID-19 pandemic.

Literature investigating the use of telehealth for the management of musculoskeletal pain is growing. Systematic reviews have demonstrated that telehealth can provide improvements in pain, physical function and disability that are similar to that of usual face-to-face care for individuals with musculoskeletal conditions such as osteoarthritis for the knee and hip. The use of telehealth also seems to increase exercise adherence for a variety of musculoskeletal conditions. To our knowledge, digital self-management programs for OA of the hand have not yet been evaluated.

Joint Academy® (JA), a digitally delivered treatment program with exercise and patient education was developed to increase access to and facilitate implementation of guideline derived and evidence-based treatment for OA. The first JA program was introduced in 2016 for persons with hip- and knee OA and participants reported reduced pain and improved function during up to 48 weeks of treatment. A recent randomised controlled trial on patients with knee OA showed that the digital program was superior to usual care. Since late 2021, a digital program for OA of the hand is also available on the platform.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years (often much older)
* Previous physical examination regarding hand symptoms
* Long-lasting hand pain where osteoarthritis is suspected l(for example joint-specific load and/or rest pain, impaired function with stiffness, decreased grip strength, clumsiness, bone roughening of joints).
* started the treatment between 2022-XX-XX to 2022-XX-XX

Exclusion Criteria:

* Pregnancy
* Tendon disease (trigger finger, tendinopathy)
* Nerve entrapment
* Arthritis
* Acute injuries (fracture and/or distortion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participats joined the programme through recommendation by their local physiotherapist (PT), occupational therapist (OT) or orthopaedic surgeon, via online advertisements and campaigns placed on search engines and social networks, or through their insurance company. A majority of included participants had a clinical diagnosis of hand osteoarthritis from a PT, OT or physician, and all had a physical visit with a healthcare provider regarding their hand OA prior to joining JA. The clinical diagnosis of OA was confirmed by a PT or OT via telephone, or if deemed necessary the patient was recommended to seek face-to-face care before inclusion in the programme.
Sampling Method: Probability Sample
Enrollment: 846 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leif Dahlberg, Professor, Study Director — Arthro Therapeutics /Joint Academy
Locations (1):
- Joint Academy, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Dreiser RL, Maheu E, Guillou GB. Sensitivity to change of the functional index for hand osteoarthritis. Osteoarthritis Cartilage. 2000;8 Suppl A:S25-8. doi: 10.1053/joca.2000.0332. PMID 11156490
- [Background] Kim SK, Jung UH, Choe JY. Functional index for hand osteoarthritis (FIHOA) is associated with pain, muscle strength, and EQ-5D in hand osteoarthritis. Adv Rheumatol. 2021 Mar 19;61(1):19. doi: 10.1186/s42358-021-00177-5. PMID 33741081
- [Derived] Walter MM, Sirard P, Nero H, Horder H, Dahlberg LE, Tveter AT, Kjeken I, Kiadaliri A. Digitally delivered education and exercises for patients with hand osteoarthritis-An observational study. Musculoskeletal Care. 2023 Dec;21(4):1154-1160. doi: 10.1002/msc.1796. Epub 2023 Jul 8. PMID 37421256

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who did not complete 3 months of treatment was excluded from the study.
Period: Overall Study
Arm/Group | Joint Academy
Started | 846
Completed | 379
Not Completed | 467
Not completed — Lost to Follow-up | 467

BASELINE CHARACTERISTICS:
Population: Participants who enrolled in the digital treatment
Groups:
- Included Participants: The participants received 3 months of the digital treatment of Joint Academy.
  Joint Academy digital treatment: The Joint Academy® (www.jointacademy.com) program for people with hand OA consists of video instructed and progressively adaptable daily exercises, patient education through text lessons, possibility for a social chat group with other patients and a continuous asynchronous chat function with a personal reg. physiotherapist who supervises the patient during the full participation period. The program also contains three telephone consultations with a physiotherapist that were compulsory, one at the start, one after six weeks and one after three months.
- Excluded Participants: Participants who enrolled to Joint Academys digital treatment but did not complete three months treatment.
  Joint Academy digital treatment: The Joint Academy® (www.jointacademy.com) program for people with hand OA consists of video instructed and progressively adaptable daily exercises, patient education through text lessons, possibility for a social chat group with other patients and a continuous asynchronous chat function with a personal reg. physiotherapist who supervises the patient during the full participation period. The program also contains three telephone consultations with a physiotherapist that were compulsory, one at the start, one after six weeks and one after three months.
- Total: Total of all reporting groups
Arm/Group | Included Participants | Excluded Participants | Total
Number analyzed (Participants) | 379 | 467 | 846
Age, Continuous [Mean (Standard Deviation); unit: years]
  All participants | 64.6 (9.3) | 62.7 (10.6) | 63.6 (10.1)
Age, Customized [Count of Participants; unit: Participants] — Population: Distribution of different age groups of participants included in the analysis (participants who completed 3 months of treatment).
  Participants
    Participants included in analysis: number analyzed (Participants) | 379 | 0 | 379
    Participants included in analysis: 28-59 years old | 108 |  | 108
    Participants included in analysis: 60-69 years old | 147 |  | 147
    Participants included in analysis: 70 years old or older | 124 |  | 124
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285 | 374 | 659
  Male | 94 | 93 | 187
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 379 | 467 | 846

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity (Numerical Rating Scale NRS, Discrete Boxes 0-10, Higher Score Mean Worse Pain)
Description: Pain intensity was assessed using the Numerical Rating Scale (NRS, discrete boxes 0-10) with the instruction: "Mark on this scale how much pain you had in your hand over the past week." The NRS ranged from 0, representing no pain, to 10, representing the maximum pain imaginable. A higher score indicated greater pain intensity.
  Participants completed mandatory self-assessment questionnaires at baseline and again at 3 months of treatment. All responses were self-reported and entered directly via the digital program interface.
Time Frame: Change in pain intensity from baseline to 3 months of treatment.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Joint Academy
Number analyzed (Participants) | 379
Units on a scale | -1.30 [-1.49 to -1.12]

2. Secondary Outcome: Functional Index for Hand OsteoArthritis (FIHOA 0 - 30 Higher Score Means Worse Outcome)
Description: The FIHOA is a 10-item questionnaire based on a semi-quantitative assessment scoring the disease on a 4-point scale with a total scoring from 0 to 30 where a higher score equals more functional impairments. The FIHOA has been shown to be valid, sensitive, clinically relevant for the population and shown consistency and acceptable reliability. The literature also suggests it is associated with pain, muscle strength and health related quality of life in people with hand OA. All outcomes were self-assessed and self-entered using the digital program interface.
Time Frame: Change of Functional Index for Hand OsteoArthritis-score between baseline to 3 months of treatment
Measure: Mean (95% Confidence Interval); unit: score on a scale. Mean change.
Arm/Group | Joint Academy
Number analyzed (Participants) | 379
score on a scale. Mean change. | -0.81 [-1.02 to -0.60]

3. Other Pre Specified Outcome: Analgesic Use
Description: Analgesic use was assessed with the question: "In the past month, have you taken any medication for the pain in your hand?" (response options: Yes or No).
  This measure represents the absolute count of participants who reported a decrease in analgesic use from baseline to the 3-month follow-up (saying Yes at baseline but No at follow up.
Time Frame: Reduction in the number of participants using analgesics from baseline to the 3-month follow-up.
Population: Not all participants answered the question regarding analgesic use.
Measure: Count of Participants; unit: Participants
Arm/Group | Joint Academy
Number analyzed (Participants) | 331
Participants | 22

4. Other Pre Specified Outcome: Willingness for Surgery
Description: Question: "Based on your symptoms, are you considering to undergo surgery of your hand?" Options: "No, I'm not; Yes, I'm considering surgery but it's not yet scheduled; Yes, surgery is scheduled; Surgery has been performed (only asked at follow up); I don't know"
  This measure represents the absolute count of participants reporting reduced willingness to undergo surgery from baseline to the 3-month follow-up.
Time Frame: Reduction in the number of participants wanting to undergo surgery from baseline to the 3-month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Joint Academy
Number analyzed (Participants) | 379
Participants | 5

5. Other Pre Specified Outcome: Fear of Physical Activity
Description: Fear of physical activity was assessed with the question: "Are you concerned that your finger joints may be damaged by physical activity or exercise?" (response options: Yes or No).
  This measure represents the absolute count of participants reporting a reduction in fear of physical activity from baseline to the 3-month follow-up.
Time Frame: Reduction in the number of participants responding "yes" from baseline to the 3-month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Joint Academy
Number analyzed (Participants) | 379
Participants | 17

6. Other Pre Specified Outcome: Stiffness in Affected Joint (NRS, 0-10, Higher Score Mean Worse Outcome)
Description: Question "Mark on the scale how much stiffness you have felt in your left/right hand due to your osteoarthritis during the past week" with a NRS ranging from 0 (none) to 10 (extreme stiffness) where a higher score equals more stiffness
Time Frame: At baseline and 3 months
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Joint Academy
Number analyzed (Participants) | 379
Units on a scale | -0.81 [-1.02 to -0.60]

7. Other Pre Specified Outcome: Received Injection at the Affected Joint (Yes/no)
Description: In the past month, have you received an injection in your "index joint" for the pain?
Time Frame: Reduction in the number of participants answering "yes" between baseline and 3 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Joint Academy
Number analyzed (Participants) | 379
Participants | 17

ADVERSE EVENTS:
Time Frame: Adverse events were not recorded
Arm/Group | Joint Academy
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT05499559/Prot_SAP_000.pdf